CLINICAL TRIAL: NCT02619526
Title: Comparative Effects of Nebivolol and Carvedilol on Diastolic Function of the Left Ventricle in the Elderly Heart Failure Patients With Preserved Ejection Fraction: Study Protocol for a Randomized Controlled Trial
Brief Title: Comparative Effects of Nebivolol and Carvedilol on Diastolic Function in the Elderly Heart Failure Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A University (Other)
Collaborators: Menarini Group (Industry)
Responsible Party: Principal Investigator, Kyungil Park, Assistant Professor, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-174
Record Dates: First submitted 2015-11-25; First posted 2015-12-02 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Nebivolol; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebivolol (Experimental): Nebivolol 10mg, once a day
  Interventions: Drug: Nebivolol
- Carvedilol (Active Comparator): Carvedilol 25mg, twice a day
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 10mg, once a day
  Arms: Nebivolol
Drug: Carvedilol — Carvedilol 25mg, twice a day
  Arms: Carvedilol

SUMMARY:
Heart failure (HF) is a common and disabling condition in the elderly. Randomized clinical trials and meta-analyses have clearly demonstrated that long-term use of β blockers improves the outcomes of patients with HF. However, limited data have been available on the treatment of HF with preserved ejection fraction (EF) in the elderly. No study has specifically compared the relative effectiveness of carvedilol and nebivolol in treating HF in old age patients with preserved EF.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, open-label, active controlled study designed to investigate effects of nebivolol and carvedilol on diastolic function of the left ventricle (LV) in the elderly HF patients with preserved EF.

Patients will be included in the study if they had LVEF ≥ 40%, NYHA functional class I, II or III, and clinical stability without hospital admission for HF in the preceding 3 months.

ELIGIBILITY:
Inclusion Criteria:

* more than 70 years
* EF ≥ 40%

Exclusion Criteria:

* contraindication to the study drug

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the ratio of transmitral E velocity to early diastolic mitral annular velocity (E/E') | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Ho Park, MD, Principal Investigator — Dong-A University
Locations (1):
- Department of Internal Medicine,Dong-A University College of Medicine, Busan, South Korea

REFERENCES:
- [Derived] Park K, Park TH. Comparative effects of nebivolol and carvedilol on left ventricular diastolic function in older heart failure patients with preserved ejection fraction: study protocol for a randomized controlled trial. Trials. 2016 Nov 3;17(1):530. doi: 10.1186/s13063-016-1656-y. PMID 27809882